CLINICAL TRIAL: NCT03851315
Title: Permanent Left Bundle Branch Area Pacing for Atrioventricular Block
Brief Title: Left Bundle Branch Area Pacing in AVB Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fu Wai Hospital, Beijing, China (Other)
Responsible Party: Principal Investigator, Fan Xiaohan, MD., PhD., Professor of Medicine, Deputy Director of Arrhythmia Center in Fuwai hospital, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: LBBAP-001
Record Dates: First submitted 2019-02-18; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Atrioventricular Block; Left Bundle Branch Area Pacing
Keywords: Atrioventricular Block; left bundle branch area pacing
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- LBBAP group: patients received left bundle branch area pacing
  Interventions: Device: permanent left bundle branch area pacing
- traditional RVP group: Age and sex-matched patients received traditional right ventricular pacing

INTERVENTIONS:
Device: permanent left bundle branch area pacing — Implant the pacing lead in the left bundle branch area instead of traditional RV pacing site(septal or apical). Successful LBBAP was defined as the paced QRS morphology of right bundle branch block pattern in lead V1 and QRS duration (QRSd) less than 130ms.
  Groups: LBBAP group

SUMMARY:
Right ventricular pacing (RVP) causes left ventricular mechanical dyssynchrony by inducing electrical interventricular and intraventricular dyssynchrony. His bundle pacing may restore the the atrioventricular, interventricular and intraventricular electrical synchronization, however, Increased pacing threshold might result in the early depletion of the pacemaker, and finally brought on pacemaker replacement, which was one of the major causes of device infection. Pacing the left bundle branch beyond the conduction block site might achieve a low and stable output and narrow QRSd. The investigators were prepared to consecutively include patients with atrioventricular block, divided into the left bundle branch area pacing(LBBAP) group and the conventional right ventricular pacing group. The electrophysiological characteristics of LBBAP and right ventricular pacing were compared with ECG characteristics. The left and right ventricular synchrony and left and right cardiac function were evaluated by 3D ultrasound, and the short-term and long-term safety and efficacy of LBBAP were evaluated.

DETAILED DESCRIPTION:
This study is intended to be included in Fuwai hospital for admission to the atrioventricular block, with permanent pacemaker implant indications recommended by current guidelines. Patients were assessed for preoperative electrocardiogram, quality of life scores, cardiac function, and left and right ventricular synchrony. Patients were followed up by regular outpatients. The electrocardiogram, quality of life score, echocardiographic function, left and right ventricular synchrony, pacing parameters and pacing ratio were evaluated immediately after surgery, 3 months, 6 months, and 12 months after surgery. At the same time, the left bundle branch area pacing success rate, complications during intraoperative and postoperative follow-up were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years old;
2. Atrioventricular block patients with indication for permanent ventricular pacing;
3. LVEF> 40%;
4. With informed consent signed

Exclusion Criteria:

1. Persistent atrial fibrillation;
2. Moderate or more severe valvular disease;
3. Hypertrophic cardiomyopathy；
4. Myocardial amyloidosis；
5. With indication for CRT or ICD implantation according to the current guideline;
6. Poor condition of the acoustic window because of emphysema or other reasons;
7. Patients refused postoperative follow-up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive AVB patients with indications for ventricular pacing according to 2013 ESC/EHRA Guidelines. Patients with persistent atrial fibrillation or indications for cardiac resynchronization therapy or implantable cardioverter defibrillator implantation , hypertrophic cardiomyopathy, myocardial amyloidosis, or refused postoperative follow-up were excluded. All patients should sign written informed consent for agreement of the implantation procedure.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
The synchronization status change at 3 months and 1 year as compared with baseline status. | 3 months and 1 year
  Left ventricualr strain change from baseline to 3 month, from baselin to 1 year post operation.

SECONDARY OUTCOMES:
Pacing threshold change at 3 months and 1 year as compared with baseline status. | 3 months and 1 year
  The pacing threshold changes between 3-month and baseline status, changes between 1 year and the baseline status.
LBBAP related adverse events at 3 months and 1 year as compared with baseline status. | 3 months and 1 year
  The adverse events includes perforation, acute myocardial infarction, loss of capture, increase of pacing threshold, et al. These events were evaluated at baseline, 3 months and 1 year after the procedure, respectively.
left ventricular ejection fraction change at 3 months and 1 year | 3 months and 1 year
  Left ventricular ejection fraction change from baseline to 3 month, from baselin to 1 year post operation.
Right ventricular ejection fraction change at 3 months and 1 year | 3 months and 1 year
  Right ventricular ejection fraction change from baseline to 3 month, from baselin to 1 year post operation.
Left ventricular end systolic diameter change at 3 months and 1 year | 3 months and 1 year
  Left ventricular end systolic diameter change from baseline to 3 month, from baselin to 1 year post operation.
Left ventricular end diastolic diameter change at 3 months and 1 year | 3 months and 1 year
  Left ventricular end diastolic diameter change from baseline to 3 month, from baselin to 1 year post operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Wai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vijayaraman P, Naperkowski A, Ellenbogen KA, Dandamudi G. Electrophysiologic Insights Into Site of Atrioventricular Block: Lessons From Permanent His Bundle Pacing. JACC Clin Electrophysiol. 2015 Dec;1(6):571-581. doi: 10.1016/j.jacep.2015.09.012. Epub 2015 Oct 17. PMID 29759411
- [Result] Huang W, Su L, Wu S, Xu L, Xiao F, Zhou X, Ellenbogen KA. A Novel Pacing Strategy With Low and Stable Output: Pacing the Left Bundle Branch Immediately Beyond the Conduction Block. Can J Cardiol. 2017 Dec;33(12):1736.e1-1736.e3. doi: 10.1016/j.cjca.2017.09.013. Epub 2017 Sep 22. PMID 29173611
- [Result] Chen K, Li Y, Dai Y, Sun Q, Luo B, Li C, Zhang S. Comparison of electrocardiogram characteristics and pacing parameters between left bundle branch pacing and right ventricular pacing in patients receiving pacemaker therapy. Europace. 2019 Apr 1;21(4):673-680. doi: 10.1093/europace/euy252. PMID 30462207
- [Result] Guo XG, Liu X, Zhou GB, Sun Q, Yang JD, Luo B, Ouyang F, Ma J, Zhang S. Clinical, electrocardiographic, and electrophysiological characteristics of left upper septal fascicular ventricular tachycardia. Europace. 2018 Apr 1;20(4):673-681. doi: 10.1093/europace/euw429. PMID 28160481
- [Result] Upadhyay GA, Cherian T, Shatz DY, Beaser AD, Aziz Z, Ozcan C, Broman MT, Nayak HM, Tung R. Intracardiac Delineation of Septal Conduction in Left Bundle-Branch Block Patterns. Circulation. 2019 Apr 16;139(16):1876-1888. doi: 10.1161/CIRCULATIONAHA.118.038648. PMID 30704273
- [Derived] Li X, Zhang J, Qiu C, Wang Z, Li H, Pang K, Yao Y, Liu Z, Xie R, Chen Y, Wu Y, Fan X. Clinical Outcomes in Patients With Left Bundle Branch Area Pacing vs. Right Ventricular Pacing for Atrioventricular Block. Front Cardiovasc Med. 2021 Jul 8;8:685253. doi: 10.3389/fcvm.2021.685253. eCollection 2021. PMID 34307499